CLINICAL TRIAL: NCT01309139
Title: An Open Label, Randomised, Two-way Crossover Phase I Study to Assess Safety, Tolerability and Pharmacokinetics of the Fixed Dose Combination of Tiotropium Plus BI 54903 Via Respimat® B Versus the Combination of the Monoproducts of Tiotropium Via Respimat® A and BI 54903 Via Respimat® B in Healthy Volunteers
Brief Title: Pharmacokinetics of the Fixed Dose Combination of Tiotropium Plus BI 54903 Versus the Combination of the Monoproducts of Tiotropium and BI 54903 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1298.2; 2010-023780-18 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-03-01; First posted 2011-03-04 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — Tiotropium Bromide

ARMS (4):
- Treatment A: Tiotropium medium dose (Experimental): Oral inhalation daily for 21 days
  Interventions: Drug: Tiotropium
- Treatment A: BI 54903 high dose (Experimental): Oral inhalation daily for 21 days
  Interventions: Drug: BI 54903
- Treatment B: Tiotropium medium dose (Experimental): Oral inhalation daily for 21 days
  Interventions: Drug: Tiotropium
- Treatment C: BI 54903 high dose (Experimental): Oral inhalation daily for 21 days
  Interventions: Drug: BI 54903

INTERVENTIONS:
Drug: Tiotropium — Medium dose of oral inhalation
  Arms: Treatment A: Tiotropium medium dose
Drug: Tiotropium — Medium dose of oral inhalation
  Arms: Treatment B: Tiotropium medium dose
Drug: BI 54903 — Medium dose of oral inhalation
  Arms: Treatment C: BI 54903 high dose
Drug: BI 54903 — Medium dose of oral inhalation
  Arms: Treatment A: BI 54903 high dose

SUMMARY:
The primary objective is to compare the systemic exposure to tiotropium and CD 1857 after treatment with the fixed dose combination (fixed dose combination (FDC), Treatment A) of tiotropium plus BI 54903 (ethanolic solution for inhalation (EIS), Respimat (RMT) B) with the systemic exposure following inhalation of the free combination (Treatment B) of tiotropium (aqueous solution for inhalation (AIS), RMT A) plus BI 54903 (EIS, RMT B), when administered once-daily over 21 days via Respimat(R) (RMT).

The secondary objectives are:

to compare the systemic exposure to tiotropium and CD 1857 after single dose administration of FDC and of the free combination of tiotropium/BI 54903 to compare the systemic exposure to BI 54903 after a single dose and at steady state after multiple doses of the FDC and of the free combination of tiotropium/BI 54903 to compare the safety and tolerability of tiotropium and BI 54903 when administered as FDC and as free dose combination, respectively

ELIGIBILITY:
Inclusion criteria:

1. Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests.
2. Age 21 to 50 years.

Exclusion criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. History or evidence of relevant psychiatric disorders or neurological disorders
5. History or evidence of relevant autonomic dysfunction (orthostatic hypotension, fainting spells or blackouts)
6. Chronic or relevant acute infections
7. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
8. Intake of any prescription drugs or over-the-counter (over the counter (OTC)) medication (vitamins, herbal supplements, dietary supplements) with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
9. Participation in another trial with an investigational drug within two months prior to administration or during the trial
10. Smoker (more than 10 cigarettes daily)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve of CD 1857 in plasma over a uniform dosing interval τ (AUCτ,ss) | on several time points until day 22
Maximum concentration of CD 1857 in plasma at steady state (Cmax,ss) | on several time points until day 22
AUCτ,ss for Tiotropium | on several time points until day 22
Cmax,ss for Tiotropium | on several time points until day 22

SECONDARY OUTCOMES:
AUCτ,ss for BI 54903 | on several time points until day 22
Cmax,ss for BI 54903 | on several time points until day 22
Ae0-24 (Amount of analyte that is eliminated in urine) for tiotropium | on Day 1 and 21
Change in physical examination | 9 weeks
Change in vital signs | 9 weeks
Change in 12-lead electrocardiogram | 9 weeks
Change in clinical laboratory tests | 9 weeks
Occurrence of Adverse Events | 9 weeks
Assessment of tolerability by the investigator | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1298.2.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany